CLINICAL TRIAL: NCT00236028
Title: A Randomized, Double-blind, Trial of Anti-TNFa Chimeric Monoclonal Antibody (Infliximab) in Combination With Methotrexate Compared With Methotrexate Alone for the Treatment of Patients With Early Rheumatoid Arthritis
Brief Title: A Safety and Efficacy Study for Infliximab (Remicade) With Methotrexate in Patients With Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003118
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Early Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of infliximab (Remicade) in patients with early rheumatoid arthritis.

DETAILED DESCRIPTION:
This is a randomized, multicenter, double-blind, active-treatment-controlled, three-arm, parallel study of chronic treatment with infliximab. This study will determine whether infliximab, at two different doses (3 mg/kg or 6 mg/kg) in combination with methotrexate (MTX), reduces the signs and symptoms (such as joint pain, swelling and stiffness) of rheumatoid arthritis. The study will also compare their effect on slowing down the joint damage associated with rheumatoid arthritis. Additional information on the safety of infliximab treatment will be obtained. The study will last for about 1 year. Patients will receive methotrexate and total of eight intravenous infusions of the study medication (Infliximab or placebo) spaced out over the first year. After the final infusion of study medication, several follow-up visits are to be made. Patients will receive methotrexate (start at 7.5mg/wk, increased to 20mg/wk by week8) and intravenous infusions of the study medication (Infliximab 3 or 6mg/kg, or placebo) at week 0, 2, and 6, and every 8 weeks thereafter through week 46.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis for at least 3 months and less than or equal to 3 years before screening
* Active disease at the time of screening and pre-infusion of the drug

Exclusion Criteria:

* Pregnant, nursing, or planning a pregnancy within 18 months of enrollment
* Incapacitated, largely or wholly bedridden, or confined to a wheelchair, or had little or no ability for self care
* Rheumatic disease other than rheumatoid arthritis or any current systemic inflammatory condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Improvement from baseline in clinical signs and symptoms, prevention of structural damage, and prevention of physical disability evaluated at week 54.

SECONDARY OUTCOMES:
Safety assessments throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Background] Visvanathan S, Wagner C, Smolen J, St Clair EW, Hegedus R, Baker D, Keenan G. IgG and IgM anticardiolipin antibodies following treatment with infliximab plus methotrexate in patients with early rheumatoid arthritis. Arthritis Rheum. 2006 Sep;54(9):2840-4. doi: 10.1002/art.22054. PMID 16948115
- [Result] Visvanathan S, Marini JC, Smolen JS, Clair EW, Pritchard C, Shergy W, Pendley C, Baker D, Bala M, Gathany T, Han J, Wagner C. Changes in biomarkers of inflammation and bone turnover and associations with clinical efficacy following infliximab plus methotrexate therapy in patients with early rheumatoid arthritis. J Rheumatol. 2007 Jul;34(7):1465-74. Epub 2007 Jun 1. PMID 17552048
- [Result] Visvanathan S, Keenan GF, Baker DG, Levinson AI, Wagner CL. Response to pneumococcal vaccine in patients with early rheumatoid arthritis receiving infliximab plus methotrexate or methotrexate alone. J Rheumatol. 2007 May;34(5):952-7. Epub 2007 Apr 15. PMID 17444589
- [Result] Smolen JS, Van Der Heijde DM, St Clair EW, Emery P, Bathon JM, Keystone E, Maini RN, Kalden JR, Schiff M, Baker D, Han C, Han J, Bala M; Active-Controlled Study of Patients Receiving Infliximab for the Treatment of Rheumatoid Arthritis of Early Onset (ASPIRE) Study Group. Predictors of joint damage in patients with early rheumatoid arthritis treated with high-dose methotrexate with or without concomitant infliximab: results from the ASPIRE trial. Arthritis Rheum. 2006 Mar;54(3):702-10. doi: 10.1002/art.21678. PMID 16508926
- [Derived] Mack ME, Hsia E, Aletaha D. Comparative Assessment of the Different American College of Rheumatology/European League Against Rheumatism Remission Definitions for Rheumatoid Arthritis for Their Use as Clinical Trial End Points. Arthritis Rheumatol. 2017 Mar;69(3):518-528. doi: 10.1002/art.39945. PMID 27696724
- See also: A Randomized, Double-blind, Trial of Anti-TNFa Chimeric Monoclonal Antibody (Infliximab) in Combination with Methotrexate Compared with Methotrexate Alone for the Treatment of Patients with Early Rheumatoid Arthritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=142&filename=CR003124_CSR.pdf